CLINICAL TRIAL: NCT06293105
Title: Responding to Homelessness, Multiple Exclusion and Stigma: Developing a Complex Public Health Intervention Approach
Brief Title: Social Responses to Stigma
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Groundswell (Unknown); Lambeth Service Users Council (Unknown); Museum of Homelessness (Unknown); Inclusive Insight (Unknown)
Responsible Party: Sponsor
Other Study IDs: MR/T040688/1
Record Dates: First submitted 2023-11-02; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Stigma, Social; Drug Use
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People who are homeless: People who are currently homeless, as per UK Government definition, or have experience of homelessness.
  Interventions: Other: Qualitative interview, participant observation
- Stakeholders: People with work or other experience relating to homelessness in London
  Interventions: Other: Qualitative interview, participant observation

INTERVENTIONS:
Other: Qualitative interview, participant observation — Qualitative in-depth interviews to explore experiences of and perspectives on stigma and discrimination, linked to being present in settings where there is participant observation

SUMMARY:
The Social Responses to Stigma study will explore experiences of stigma and discrimination amongst people who are homeless in south London, and then seek to understand how this stigma is created, mediated or mitigated within health, social, housing and legal care and support systems and social contexts.

The methodology is an ethnographic case study of the south London care and support system and its social context. The study will use a range of methods for data collection: interviews with people who are homeless, delivery stakeholders, and policy makers; a survey of peoples' experiences; observation within selected care sites; and gathering of documentary sources.

The study will be implemented through two parallel studies. The first, with KCL-REMAS approval, will operate in non-NHS sites. The second, with NHS-IRAS approval, will operate in NHS sites. The protocols are aligned with adaptations for each type of site.

A linked method to develop theory is cross-case comparison between South London and Vancouver, Canada, through secondary data analysis to linked studies ongoing there. The study will be ongoing from 2022 until January 2025. The project is funded in two phases, with potential to extend the study by a further three years, to January 2028.

The results of the study will inform the design of a novel intervention strategy to address the social dimensions of stigma. Subject to additional funding applications, the intervention strategy will be piloted and evaluated from 2025 onwards. The study results will be disseminated through scientific publications, public reports and a range of public and policy engagement activities.

DETAILED DESCRIPTION:
Background Stigma refers to people being 'marked' in society's eyes as lesser, unworthy or disgraced, and then consequently experiencing discrimination. This stigma that often focuses on people who are homeless, and how that intersects with drug use, mental health and other identities and experiences, is widely understood as a cause of ill-health through being a persistent barrier to accessing support and services and through creating conditions and experiences that deny or limit the determinants of health.

Stigma scholarship increasingly emphasises the role of care systems and social context in producing stigma. Numerous studies have drawn attention to how stigma is experienced within health care settings. There is in turn a wide literature exploring how systems of criminalisation of drugs or regimes of welfare benefits can be understood to generate stigma. In consequence, stigma can be understood as a phenomena experienced across different settings and that emerges from long-running structural processes.

Rationale for the study Whilst there is increasing understanding of the social aspects of stigma and their complexity, theory that delineates specific pathways by which particular experiences relate to social factors is still limited. Indeed, social theory on stigma can be characterised as having a 'gap': understanding of micro-scale interactions is rich, and there is increasing analysis of macro-scale influences, but little understanding of how these levels interact. In the absence of such theory there is little to guide empirical research and then public health interventions that could address these dimensions of stigma.

Corresponding to the social theory gap, interventions to address stigma at a social level are limited. Current evidence indicates short-term impact from individual and inter-personal level interventions to prevent stigma in health care settings, but little progress in developing interventions seeking coordinated change at multiple levels. Stigma scholars and policymakers agree that we need new theory, interventions and evaluation methods to respond to the systemic nature of stigma.

Overlapping with the specific debate on stigma, public health is increasingly seeking to develop 'complex systems interventions', which could provide a route to thinking of how to respond to the social roots of stigma. A complex system intervention approach could seek change across multiple overlapping systems to enable, in combination, access to care, social support and housing, and consequently significant impact on health and welfare.

Theoretical framework The need to further develop theory to understand the social processes involved in stigma to in turn inform complex systems level interventions could be addressed by the application of social practice theory.

Social practice theories are prominent in social science, but under-developed in their application to public health intervention. Furthermore, social practice theory is little used with respect to studying stigma, despite the overlapping concern for power, inequalities and how concepts of symbolic violence have considerable analytical value for understanding stigma.

A central contention of the Social Responses to Stigma project is that greater integration of the literatures on social practice theory and then stigma could bring powerful insights.

Research questions and aims The Social Responses to Stigma project aims to address the theoretical gap on stigma theory and the need for novel interventions addressing the social causes of stigma. The project will specifically develop the application of social practice theory to stigma, and through this theorise a novel system level intervention addressing the stigma experienced by people who are homeless. The outcome sought by the project is a reduction in the forms of stigma that complicate homelessness and associated ill-health.

The project is funded by a UKRI Fellowship and has two phases. The first phase, with funding awarded, years 1-4 (Feb 2021 to Jan 2025) will theorise and empirically study stigma as it relates to homelessness in south London; the study described in this protocol is a core part of this first phase of the fellowship. Linked work in the first phase will involve comparative analysis to research in Canada, and then a multi-stakeholder process to co-produce a novel intervention strategy that addresses the social causes of stigma.

A second phase, with funding contingent on an extension application, in years 5-7, will implement and evaluate the novel strategy within London, and then explore the application of the intervention approach in other settings, in the UK and globally.

The study described in this protocol has four work packages: WP1 is an ethnographic study of stigma and how it is experienced and generated within the care systems of south London; WP2 will further generate the theory developed through WP1 through comparative analysis to linked studies in Canada; WP3 will focus on developing a novel intervention strategy through a multi-stakeholder process in south London; WP4 will seek ongoing public and stakeholder engagement in the study to ensure its relevance and utility.

WP 1 objectives and research questions Objective 1.1 - to develop a typology describing how stigma is experienced by people who are homeless in south London RQ1.1.1 how do people who are homeless experience stigma (anticipated, enacted, internalised)? RQ1.1.2 how are these experiences located in different elements of the south London care and support system? RQ1.1.3 how do these experiences relate to intersections of homelessness with drug use (both controlled drugs and alcohol), mental health status, gender, migration, race and ethnicity, sexuality, and HIV status? RQ1.1.4 what are the impacts on health and welfare of these experiences of stigma and discrimination?

Objective 1.2 - to analyse the forms of stigma described in objective 1.1 in relation to the system and social setting of south London, using Bourdieu's social practice theory RQ1.2.1 How are the experiences of stigma described in obj 1.1 embedded in everyday practices that either produce or manage them? A - what are the fields in which these practices occur? B - who are the actors involved in the stigma described, and what are the relations between them, and what position do they occupy in the system? C - what is the habitus associated with each (group of) actors?

Objective 1.3 - to explore change, or potential for it, in the stigma and stigma practices described in Obj 1.1 and 1.2, using Bourdieu's social practice theory RQ1.3.1 how might the habitus, fields and capitals involved in producing stigma practices change? RQ1.3.2 what are the contributions of particular existing interventions to changing habitus, fields and capitals? Considering in particular: peer-led or peer-involved services, community driven initiatives andhealth system leadership.

WP2 objectives Objective 2.1 to refine theory from WP1, with particular emphasis on the role of the criminalisation of drugs in producing stigma RQ2.1.1 how do different regimes of drug criminalisation shape experiences of stigma and discrimination amongst people who are homeless?

WP3 objectives Objective 3.1 produce an analysis of stigma in south London, in the context of existing evidence for stigma and related interventions, to guide stakeholder consultations Objective 3.2 implement a multiple stakeholder process to co-develop a complex systems intervention strategy to address stigma

WP4 objectives Objective 4.1 ensure a range of stakeholders - including people who are homeless, policy makers, service delivery professionals, and members of the public - are engaged in ongoing plans for data collection and results from analysis to ensure relevance of study findings and outputs

Study design and methods of data collection and analysis An ethnographic approach will develop a case study of stigma in south London, implemented with a participatory and applied orientation.

Ethnography Ethnographic research aims to understand phenomena as they are experienced and have meaning for people, and to do this through sustained and immersive presence in a research setting. Through sustained presence in settings where stigma is experienced and created, and using a combination of methods of observation, interviews and documentary sources, the study will engage with how stigma is experienced and the contexts involved the aim is not necessarily to observe discrimination in practice, but of the contexts for it, and especially how stigma is conceptualised as a dispersed and multi-dimensional phenomena. The study will study these multiple dimensions, and through theoretically driven analysis building on social practice theory explore how they combine to produce the experiences seen.

Case study of the south London care and support system The ethnography will develop a case study of stigma and how it is produced and managed within the south London care and support system. The 'case' is the south London care and support system, comprising health and social care and other services or official institutions which people who are homeless engage with; which includes, but is not limited to: health care, housing services, welfare services, policing and criminal justice. This selection of the case is a response to the proposition that stigma is produced and enacted within, or mediated by, a particular system, reflecting an effort to understand how different components of the system interact (e.g. health care and housing services), and then in turn how this same system is intended as a priority for the consequent public health intervention. Within the 'case' of the south London care and support system the study will in turn study a range of 'sub-cases' or embedded units of analysis - e.g. individual hospitals, or hostels and day centres.

The case of the system of care and support is then understood as embedded within the 'context' of south London, and how that in turn is situated with London and then the UK. Through engaging with 'context' - such as national and international policy that criminalises drug use - the study will explore how different factors combine to create local manifestation of stigma, and also then assist in understanding how findings for the specific case of south London may relate to other settings.

The case study will be the basis for theorising how stigma is produced, enacted and managed within this particular system and social setting, through exploring how the case relates to other similar situations, with this shaped by understanding the relations to context, and also in terms of how internal comparison within the case - e.g. comparing different embedded units of analysis, such as hostels - can aid in theorising causation of particular processes. Theorising and analytical generalisability will also be supported through cross-case comparison between the study in London and then existing data sets from other studies in Vancouver (See work package 2). Analytical generalisation will also be supported by small-scale data collection in different cases or sub-cases (e.g. hostels in other parts of London, or other cities in the UK) to explore how comparable the experiences described are.

ELIGIBILITY:
People who are homeless

Inclusion Criteria:

Homelessness, in line with UK Government definitions, will be understood in an expansive way, to include past or current experiences of:

* People who are rough sleeping (meaning people without homes who sleep outside or somewhere not designed for habitation)
* people who are temporary residents of hostel accommodation (such as emergency night shelters, short-stay hostels, longer stay hostels, domestic violence safe houses, safe houses for victims of modern slavery and probation hostels)
* people who are in unsupported temporary accommodation (such as B&Bs), People who use day centres that provide support (such as food, showers, clothing and advice) for people experiencing homelessness
* People staying temporarily with family and friends ('sofa surfing'), and
* people with a history of homelessness (as defined by the groups above) who are at high risk of becoming homeless again because of ongoing complex health and social care needs.

The study will include people over the age of 18 (and exclude those under this), and with no upper age limited.

Participants would be principally based in, or frequently spend time in, the three boroughs of Lambeth, Lewisham and Southwark. Reflecting the effort to explore analytical generalisability of findings, the study may also include people with experience of homelessness beyond the three boroughs (but would still need to have experience, and be aged over 18).

Exclusion Criteria:

* Unable to give informed consent

Stakeholders Stakeholders are defined as individuals 1) working in care and support services, or services that engage people who are homeless, and whether that is in delivery, planning or management of these, or 2) with experience or position that gives insight to processes of care and support, engagement or in stigma itself. This will include staff working across health, welfare and judicial settings, including providers as well as administrative and reception staff in these settings. Those involved in policy, such as commissioners, councillors will also be included. We will also include community activists, family members and others otherwise actively engaged in issues relating to homelessness as stakeholders.

The study will include people over the age of 18 (and exclude those under this), and with no upper age limited.

Participants would be principally based in, or frequently spend time in, the three boroughs of Lambeth, Lewisham and Southwark. Reflecting the effort to explore analytical generalisability of findings, we may also include stakeholders beyond the three boroughs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population is derived from people using or working in services relating to homelessness and health in south London.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Experiences of stigma and discrimination | 2022-2025
  The outcome the study is focused on is describing peoples' experiences of stigma and discrimination. As an ethnographic study there isn't a 'primary outcome' in the statistical sense of the term, that will use a scale. Instead, the study is aiming to identify experiences of stigma and discrimination and then qualitatively explore their system context.

CONTACTS AND LOCATIONS:
Locations (1):
- to Be Determined, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No